CLINICAL TRIAL: NCT01830478
Title: Phase II Study of Lenalidomide in Combination With Rituximab (R) for the Treatment of Indolent Non Follicular Non Hodgkin Lymphoma (NHL).
Brief Title: Lenalidomide Plus Rituximab (R) in Non Follicular NHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFL08
Record Dates: First submitted 2013-04-05; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Indolent Non Hodgkin Lymphoma
MeSH Terms: interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide and Rituximab (Experimental): Lenalidomide 20 mg once daily on days 1-21 of 28 days cycle for up to 6 courses and Rituximab 375 mg/m2 at day 14 of every course.
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 20 mg p.o. once daily, days 1-21 every 28 days, for 6 cycles
  Other Names: Revlimid
Drug: Rituximab — Rituximab 375 mg/m2 intravenously, day 14 of every course for 6 cycles
  Other Names: Mabthera

SUMMARY:
The purpose of this study is to determine whether lenalidomide in association with rituximab is effective in the treatment of patients with indolent non follicular NHL relapsed after >=2, but less than 4 prior lines of (immuno)chemotherapy.

DETAILED DESCRIPTION:
Single arm, multicenter, open-label study divided in two phases: 1. Induction phase; 2. Follow-up phase. Enrolled patients will start the induction phase and receive the courses of R-Lenalidomide. At the end of the third cycle of R-Lenalidomide (week 12 of the study), the patients will be evaluated for tumor response (complete assessment); the patients with Progressive Disease (PD) will be withdrawn of the study. Two weeks after the end last courses of R-Lenalidomide (week 26 of the study) patients will be evaluated for tumor response (complete assessment). Patients with Complete Response (CR) and Partial Response (PR), and with a stable disease will undergo the follow up phase, while patients with PD will be withdrawn of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed diagnosis of B-Cell non follicular NHL according to REAL/WHO Classification: small lymphocytic lymphoma, lymphoplasmacytic lymphoma/Waldenstrom macroglobulinemia, nodal marginal zone lymphoma, splenic marginal zone lymphoma, extranodal non-gastric marginal zone lymphoma
* Availability of tissue biopsy mandatory when suspected pathological sites (nodal or extranodal) are easily accessible and in presence of extranodal non-gastric marginal or nodal marginal zone lymphoma diagnosis. In the other cases bone marrow biopsy, when representative, may be considered sufficient for defining lymphoma histotype
* Disease relapsing after >=2, but less than 4 prior lines of (immuno)chemotherapy. At least one of previous treatment had to include rituximab
* Presence of at least one of the following criteria for the definition of active disease: systemic symptoms, bulky disease, progressive marrow failure and/or splenomegaly and/or lymph adenopathy
* Age 18-75
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group (ECOG) <=2
* Left ventricular ejection fraction (LVEF) >=45%
* Creatinine clearance >= 50 mL/min calculated by Cockcroft-Gault estimation; patients with creatinine clearance >= 30 and < 50 mL/min, at physician discretion could enter the study starting at lenalidomide dose level -2 (10 mg)
* Total bilirubin up to 2 x upper limit of normal(ULN). Total bilirubin values higher than 2 x ULN are admitted if related to localization of the disease
* Alkaline phosphatase up to 2 x ULN and transaminases up to 3 x ULN
* Female and male patients must agree to participate in pregnancy prevention program signing informed Consent (paragraph 5.4.)
* Written informed Consent

Exclusion Criteria:

* Previously untreated patients
* Patients with diagnosis of typical Chronic Lymphocytic Leukemia (CLL)
* Women and men not agreeing to take adequate contraceptive precautions during and for at least 4 weeks after cessation of therapy
* Pregnant or lactating women
* History of other malignancies within 3 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer, low grade, early stage localized prostate cancer treated surgically with curative intent, good prognosis ductal carcinoma in situ (DCIS) of the breast treated with lumpectomy alone with curative intent
* Active bacterial, viral or fungal infection requiring systemic therapy
* Concurrent co-morbid medical condition which might exclude administration of therapy
* Cardiac insufficiency (NYHA grade III/IV)
* Myocardial infarction within 6 months of entry on the study
* Severe chronic obstructive pulmonary disease with hypoxemia
* Severe diabetes mellitus difficult to control with adequate insulin therapy
* Hypertension that is difficult to control
* Creatinine clearance < 30 mL/min calculated by Cockcroft-Gault estimation
* Absolute neutrophil count (ANC) <= 1 x 109/L, unless due to lymphoma involvement and not responding to 5 days of Granulocyte colony-stimulating factor (G-CFS) treatment
* Platelets count <=75.000/mm3, unless due to lymphoma involvement
* HIV and Hepatitis B virus (HBV) positivity
* Hepatitis C virus (HCV) positivity in presence of high level of virus replication and Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) > x 2.5 ULN
* Central nervous system (CNS) involvement by lymphoma
* Known hypersensitivity or anaphylactic reactions to murine antibodies or proteins
* Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy | Two weeks after the completion of Rituximab + Lenalidomide
  Evaluate the efficacy in term of Overall Response Rate (Complete Response + Partial Response) and Tumour Control Rate (Complete Response + Partial Response + Stable Disease)

SECONDARY OUTCOMES:
Assess the safety | From start of treatment for all follow up period (18 months)
  The safety will be evaluated on the basis of recorded toxicities graded on a scale of 1 to 5 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Sacchi, MD, Principal Investigator — Gruppo Italiano Studi Linfomi
Locations (1):
- Centro Oncologico Modenese, Modena, MO, Italy